CLINICAL TRIAL: NCT00018824
Title: The Treatment of Late Life Major Depression Complication by Alcohol
Brief Title: Treating Alcohol Use In Older Adults With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Oslin, David - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBS-009-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Alcoholism; Depression
MeSH Terms: conditions — Alcoholism; Depression | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Naltrexone
  Interventions: Drug: NALTREXONE
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NALTREXONE
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to test the efficacy combining a treatment for depression with a treatment for alcohol dependence.

DETAILED DESCRIPTION:
This study aims to study 80 patients with comorbid alcohol dependence and a depressive syndrome. After appropriate detoxification, patients are started on either naltrexone 50 mg or placebo. After one week, sertraline is added in an open label fashion. It is hypothesized that those patients receiving combination therapy will last 3 months with follow-up tracking lasting 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 55
* Current depressive syndrome
* Current alcohol dependence
* No psychosis
* No opioid or cocaine abuse or dependence

Exclusion Criteria:

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 1999-10; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Alcohol use' | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Oslin DW. Treatment of late-life depression complicated by alcohol dependence. Am J Geriatr Psychiatry. 2005 Jun;13(6):491-500. doi: 10.1176/appi.ajgp.13.6.491. PMID 15956269